CLINICAL TRIAL: NCT01031459
Title: An Observational 20-year, Cross-sectional, Long-term Follow up of the Patient Cohort Enrolled in the Pivotal Study of Betaseron® (Interferon Beta-1b) in Relapsing-remitting Multiple Sclerosis
Brief Title: Telephone Interview of Patients That Participated in the the Pivotal Betaferon MS Trial.
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Therapeutic Area Head, Bayer Healthcare Phamaceuticals Inc.
Other Study IDs: 14261; 20Y-LTF (Other: company internal)
Record Dates: First submitted 2009-12-08; First posted 2009-12-14 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Betaseron (Interferon beta-1b, BAY86-5046)

INTERVENTIONS:
Drug: Betaseron (Interferon beta-1b, BAY86-5046) — Telephone survey of all patients.

SUMMARY:
The purpose of this study is to investigate the clinical status of patients who participated in the original pivotal Betaseron study at 20 years after randomized treatment initiationStudy end-points include:

1. Mortality - All-cause mortality - Cause specific mortality - Multiple sclerosis-related mortality
2. EDSS (Expanded Disability Status Scale)
3. Cognition
4. Resource use
5. SPMS (Secondary Progressive Multiple Sclerosis) status
6. Employment history

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in the Betaseron pivotal study protocols TB01-35686 in the US and TB01-35886 in Canada (total, N=372)
* Patient, caregiver, or legal guardian must provide written informed consent
* Patient must confirm her/his ability and agreement to participate in the study at the beginning of the phone call

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MS that participated in the 16Y-LTF and Pivitol studies
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Descriptive exploration of mortality, EDSS, cognition, resource use, SPMS status and employment history by length of exposure to Betaseron and stratified by the original clinical trial group assignment (1.6 MIU, 8 MIU, placebo) | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (6):
  - Birmingham, Alabama
  - Tucson, Arizona
  - San Francisco, California
  - Chicago, Illinois
  - Baltimore, Maryland
  - Philadelphia, Pennsylvania
- Canada (3):
  - Vancouver, British Columbia
  - London, Ontario
  - Montreal, Quebec